CLINICAL TRIAL: NCT00349843
Title: Investigation of Multi-Purpose Solution-Based Corneal Staining and Ocular Comfort With Daily Wear FDA Group IV Hydrogel Lenses
Brief Title: Investigation of Multi-Purpose Solution-Based Corneal Staining and Ocular Comfort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P/211/04/L
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

INTERVENTIONS:
Device: Soft contact lens
Drug: Marketed soft lens multipurpose disinfection regimen

SUMMARY:
The primary objective of this study is to compare subjective ocular symptoms and corneal staining over time in a group of individuals who wear soft contact lenses on a daily wear basis, whilst they sequentially use two different contact lens care regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Agrees to wear the study lenses on a daily wear basis without the use of ocular lubricants.
2. Has an up to date pair of glasses and is willing to wear these glasses at different times during the study.
3. Is correctable to a visual acuity of 6/6 or better with their habitual correction.
4. Is willing and able to follow product usage instructions and maintain the visit schedule.
5. Is at least 18 years of age and has full legal capacity to volunteer.
6. Can be successfully fitted with study lens type.
7. Has read, understood and signed an Information Consent Letter.
8. Has a distance contact lens prescription is between -0.50 D and -9.00 D
9. Has astigmatism of ≤ 1.00 D Cyl
10. Has normal binocular vision, i.e. no strabismus, no amblyopia, and anisometropia of ≤ 1.00D
11. Has no systemic disease affecting ocular health.
12. Is not using any systemic or topical medications that will affect ocular health, accommodative function, or the ocular physiological response to the contact lenses.
13. Has clear corneas and no active ocular disease.
14. Has no known ocular or systemic allergies, which could interfere with contact lens wear.
15. Has no lid or conjunctival abnormalities, neovascularization, limbal injection, bulbar injection or corneal staining, which in the investigator's opinion is clinically significant.
16. Has not worn rigid contact lenses in the last 30 days or has corneal distortion resulting from rigid lens wear.
17. Has not worn extended wear contact lenses in the last 30 days.
18. Has had an oculo-visual examination in the last two years

Exclusion Criteria:

1. Has any active ocular disease.
2. Has any lid or conjunctival abnormalities that may, in the opinion of the investigator, interfere with the wear of contact lenses.
3. Has edema, staining, clinically significant corneal opacity, dystrophy, vascularization or iritis as viewed by slit lamp. (Trace or grade 1 equivalent limbal and bulbar injection or corneal staining is permissible at the discretion of the investigator.)
4. Is using ocular lubricants or contact lens rewetting drops on a regular basis (at least once per day)
5. Is using topical ocular prescription or any topical over-the-counter medication.
6. Is actively involved in any other research/clinical study.
7. Has worn rigid lenses or soft lenses on an extended wear basis within the last 30 days.
8. Has had corneal refractive surgery.
9. Has known sensitivity to any of the study solutions.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06

PRIMARY OUTCOMES:
The primary objective of this study is to compare corneal staining over time in
a group of individuals who wear soft contact lenses on a daily wear basis,
whilst they sequentially use two different contact lens care regimens.

SECONDARY OUTCOMES:
The secondary objective of this study is to compare subjective ocular symptoms
over time in a group of individuals who wear soft contact lenses on a daily wear
basis, whilst they sequentially use two different contact lens care regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Woods, PhD, Principal Investigator — University of Waterloo; Desmond Fonn, MOptom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada